CLINICAL TRIAL: NCT03781037
Title: Targeting Burdensomeness Among Clinic Referred Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1F31MH116603 (NIH)
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Perceived Burdensomeness Toward Others

STUDY DESIGN:
Intervention Model Description: open label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GIVE module (Experimental): The GIVE module consists of one 50-minute treatment session and a second partial session (15-20 minutes) embedded within a larger cognitive behavioral treatment (CBT) protocol for anxiety or depression. The GIVE module uses cognitive behavioral principles to target youth's beliefs that they are a burden or drain on others.
  Interventions: Behavioral: GIVE Module

INTERVENTIONS:
Behavioral: GIVE Module — The GIVE Module is a brief cognitive behavioral intervention targeting youths' beliefs that they are a burden or drain on others. It consists of two sessions embedded within a larger CBT protocol for anxiety or depression.

SUMMARY:
This study will develop and pilot test a novel intervention module targeting perceived burdensomeness toward others in 30 clinic referred youths who experience anxiety or depression and elevated levels of burdensomeness. All participants will be assigned to receive the intervention in this open trial.

DETAILED DESCRIPTION:
Suicidal ideation is prevalent and impairing in youth, with approximately 15% of high school students reporting seriously considering a suicide attempt and making a specific plan for suicide in the past 12 months. Substantial evidence documents perceived burdensomeness towards others, or the belief that one is a burden or drain on others, as a risk factor for suicide ideation in youth. This evidence highlights the potential promise of perceived burdensomeness as a novel intervention target to prevent suicide ideation in youth. The current study will develop and preliminary evaluate a novel, brief behavioral treatment module targeting perceived burdensomeness in youth that can be embedded within existing psychosocial treatments. The study will use an open trial design. The first aim of this proposal is to develop a novel, brief psychosocial intervention module (the GIVE module) targeting perceived burdensomeness towards others that can be embedded within existing CBT protocols for youth internalizing problems. The second aim is to collect data relevant to client satisfaction and reductions in perceived burdensomeness. Participants will be N=30 clinic-referred youth ages 10 to 17 years with anxiety or depressive disorders in a university-based research clinic, who display elevated levels of perceived burdensomeness. In the context on ongoing CBT for anxiety or depression, participants will complete the GIVE module at sessions 6 and 7 of the CBT protocol. It is hypothesized that perceived burdensomeness will be significantly lower after the GIVE module is administered, and that client satisfaction will be high. Data collected in this study will provide the foundation for a subsequent randomized controlled trial of the GIVE module.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of an anxiety disorder, persistent depressive disorder, or major depressive disorder
* Score > 4 on the youth self-report Interpersonal Needs Questionnaire- Perceived Burdensomeness Scale

Exclusion Criteria:

* Clinical diagnosis of a Psychotic Disorder, Autism Spectrum Disorder or Intellectual Disability
* Show high risk of imminent self-injurious behaviors
* Be involved currently in another behavioral treatment
* Not live with a primary caregiver who is legally able to give consent for the youth's participation
* Be a victim of previously undisclosed abuse requiring investigation or ongoing supervision by the Department of Children and Families.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University Center for Children and Families, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Give Module: All participants were assigned to the Give Module, consisting of one 50-minute treatment session and a second partial session (15-20 minutes) embedded within a larger cognitive behavioral treatment (CBT) protocol for anxiety or depression. The GIVE module uses cognitive behavioral principles to target youth's beliefs that they are a burden or drain on others.
Period: Overall Study
Arm/Group | Give Module
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GIVE Module
Number analyzed (Participants) | 18
Age, Customized [Count of Participants; unit: Participants]
  Between 10 and 17 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: 6-item Youth Perceived Burdensomeness Subscale of the Interpersonal Needs Questionnaire
Description: Youth self-ratings on perceived burdensomeness over the past week. Each item is scored 1-7 (1 = not at all true for me; 7 = very true for me), yielding a total between 6 and 42. Higher scores indicate higher levels of perceived burdensomeness (worse outcome).
Time Frame: post-intervention (within one week of completing the GIVE Module)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Give Module
Number analyzed (Participants) | 18
score on a scale | 9.0 (9.2)

2. Secondary Outcome: 10-item Youth Rated Warmth Subscale of the Child Report of Parental Behavior Inventory
Description: Youth ratings on parental warmth over the past week. Each of 10 items is scored 1-3 (1 = not like parent; 3 = a lot like parent), yielding a total score of 10 to 30. Higher scores indicate higher levels of parental warmth (better outcome).
Time Frame: post-intervention (within one week of completing the GIVE Module)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GIVE Module
Number analyzed (Participants) | 18
score on a scale | 13.00 (4.06)

3. Secondary Outcome: 10-item Parent Rated Warmth Subscale of the Parent Report of Parental Behavior Inventory
Description: Parent self-ratings on parental warmth over the past week. Each of 10 items is scored 1-3 (1 = not like me; 3 = a lot like me), yielding a total score of 10 to 30. Higher scores indicate higher levels of parental warmth (better outcome).
Time Frame: post-intervention (within one week of completing the GIVE Module)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GIVE Module
Number analyzed (Participants) | 18
score on a scale | 16.8 (2.8)

4. Secondary Outcome: 41-item Youth Rated Screen for Child Anxiety Related Emotional Disorders
Description: Youth self-ratings on anxiety symptom severity. Each item is scored 0-2 (0 = not true; 2 = very true), yielding a total score of 0 to 82. Higher scores indicate higher levels of anxiety (worse outcome).
Time Frame: post-intervention (within one week of completing the GIVE Module)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GIVE Module
Number analyzed (Participants) | 18
score on a scale | 43.27 (13.94)

5. Secondary Outcome: 41-item Parent Rated Screen for Child Anxiety Related Emotional Disorders
Description: Parent ratings on youth anxiety symptom severity. Each item is scored 0-2 (0 = not true; 2 = very true), yielding a total score of 0 to 82. Higher scores indicate higher levels of anxiety (worse outcome).
Time Frame: post-intervention (within one week of completing the GIVE Module)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GIVE Module
Number analyzed (Participants) | 18
score on a scale | 30.6 (14.43)

6. Secondary Outcome: 28-item Youth-rated Children's Depression Inventory - 2
Description: Youth self-ratings on depressive symptom severity. Each item is scored 0-2, yielding total scores of 0 to 56, with higher scores corresponding to more severe symptoms.
Time Frame: post-intervention (within one week of completing the GIVE Module)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GIVE Module
Number analyzed (Participants) | 18
score on a scale | 18.3 (9.6)

7. Secondary Outcome: 17-item Parent Rated Children's Depression Inventory - 2
Description: Parent ratings on youth depressive symptom severity. Each item is scored 0-3, yielding total scores of 0 to 51, with higher scores corresponding to more severe symptoms.
Time Frame: post-intervention (within one week of completing the GIVE Module)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GIVE Module
Number analyzed (Participants) | 18
score on a scale | 15.9 (8.7)

8. Secondary Outcome: 8-item Youth Rated Client Satisfaction Questionnaire
Description: Youth ratings of satisfaction with the GIVE module. Each item is score 1-4 (1 = quite dissatisfied; 4 = very satisfied), yielding total scores of 8-32. Higher scores indicate higher satisfaction (better outcome).
Time Frame: post-intervention (within one week of completing the GIVE Module)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GIVE Module
Number analyzed (Participants) | 18
score on a scale | 28.27 (2.37)

9. Secondary Outcome: 8-item Parent Rated Client Satisfaction Questionnaire
Description: Parent ratings of satisfaction with the GIVE module. Each item is score 1-4 (1 = quite dissatisfied; 4 = very satisfied), yielding total scores of 8-32.
Time Frame: post-intervention (within one week of completing the GIVE Module)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: through study completion, up to 14 weeks for each participant
Description: This intervention conferred minimal risk to participants. All participants were young (10 to 17 years) and and no study procedures put participants at risk for serious adverse events, mortality, or other adverse events.
Arm/Group | Give Module
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT03781037/Prot_SAP_000.pdf